CLINICAL TRIAL: NCT02348710
Title: Exercise Outcome Expectations Among Breast Cancer Survivors
Brief Title: Exercise Intervention for Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: Pro00059469
Record Dates: First submitted 2015-01-23; First posted 2015-01-28 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2016-08

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- exercise outcome expectation workbook (Experimental): Intervention arm participants will receive: 1) the ACS exercise and diet guidelines; and 2) an exercise outcome expectation workbook. The workbook contains self-directed activities to increase OE importance, certainty, and accessibility. The workbook will aim to make participants aware of the breadth and depth of OEs by first providing a global overview of the many positive exercise outcomes breast cancer survivors may experience. Importance will be increased through elaboration of why outcomes are important to the participant; and certainty will be increased by narrative messages from other breast cancer survivors and an oncologist. Accessibility will be increased by having the participant think about the association between exercise and its outcomes.
  Interventions: Behavioral: Exercise OE workbook
- diet workbook (Active Comparator): Attention control participants will receive via mail 1) the ACS exercise and diet guidelines; and 2) a diet workbook. The diet workbook contains the same activities as the exercise outcome expectation workbook but is focused on diet instead of exercise.
  Interventions: Behavioral: Diet workbook

INTERVENTIONS:
Behavioral: Exercise OE workbook — The workbook will aim to make participants aware of the breadth and depth of OEs by first providing a global overview of the many and diverse positive outcomes breast cancer survivors may experience. Participants will then be asked to focus on the three OEs they would most like to experience. Each section of the OE guide contains activities to target specific OE dimensions. Importance will be increased through elaboration of why outcomes are important to the participant; and certainty will be increased by narrative messages from other breast cancer survivors and an oncologist. Accessibility will be increased by having the participant think about the association between exercise and its outcomes
  Arms: exercise outcome expectation workbook
Behavioral: Diet workbook — The workbook will contain the same activities as the intervention workbook but be focused on diet instead of exercise.
  Arms: diet workbook

SUMMARY:
This randomized controlled trial will test a multicomponent intervention to increase exercise Outcome Expectations (OEs) and assess effects of OE changes on exercise intentions and levels of exercise. Sixty early stage breast cancer survivors will be recruited from the Duke Cancer Institute. Participants will be randomized to the exercise OE intervention or an attention control group. Both groups will receive the American Cancer Society diet and exercise guidelines and an accelerometer. The intervention group will also receive an OE workbook containing self-directed activities to increase OEs by focusing on OE importance (value placed on the outcome(s)), certainty (perceived probability outcome(s) will occur); and accessibility (frequency with which the outcome(s) are thought of). The attention control group will receive a workbook containing the same activities focused on diet, rather than exercise.

DETAILED DESCRIPTION:
This study will test a theory-based intervention to increase levels of exercise among breast cancer survivors, in order to help them self-manage their long-term treatment side effects. The study focuses on outcome expectations (OEs), a significant yet understudied construct that is central to most behavior change theories. OEs refer to what people expect to obtain or avoid by engaging in a behavior; thus, people exercise because they believe it will produce desired outcomes. This randomized controlled trial will test a multicomponent intervention to increase exercise OEs and assess effects of OE changes on exercise intentions and levels of exercise. Sixty early stage (IA to IIB) inactive breast cancer survivors will be recruited from the Duke Cancer Institute. Participants will be randomized to the exercise OE intervention or an attention control group. Both groups will receive the American Cancer Society diet and exercise guidelines and an accelerometer. The intervention group will also receive an OE workbook containing self-directed activities to increase OEs by focusing on OE importance (value placed on the outcome(s)), certainty (perceived probability outcome(s) will occur); and accessibility (frequency with which the outcome(s) are thought of). The attention control group will receive a workbook containing the same activities focused on diet, rather than exercise. OE importance, OE certainty, OE accessibility, exercise intentions, exercise, and self-efficacy (a potential co-variate) will be assessed through online surveys at baseline, 4-, 8-, and 12-weeks post-intervention. At each time point, accelerometer data will be collected as an objective exercise measure. Specific aims of the study are to: (1) examine trajectories of OE importance, certainty and accessibility between participants in the OE intervention arm compared to participants in the attention control arm, across four time points: baseline, 4-, 8- and 12-weeks post-intervention; and (2) examine trajectories of exercise intentions and total weekly minutes of exercise, between participants in the OE intervention arm compared to participants in the attention control arm, across four time points: baseline, 4, 8 and 12 weeks post-intervention. If the intervention increases exercise among breast cancer survivors it may lead to improved survivorship duration and quality of life. The intervention can be implemented readily in clinic settings to support survivors to exercise more and thus experience better long-term outcomes. This study also provides a foundation for a developing a nurse scientist's program of research focused on designing theory-based exercise interventions for chronically ill populations.

ELIGIBILITY:
Inclusion Criteria:

1. stage 1A - 2B breast cancer diagnosis;
2. 2 months - 10 years status post surgery, radiation and chemotherapy;
3. inactive (self-reported ≤ 150 min/wk moderate - strenuous-intensity exercise);
4. no evidence of cancer recurrence;
5. no pre-existing medical condition(s) that preclude adherence to an unsupervised exercise program (e.g., severe orthopedic conditions, scheduled hip or knee replacement within 6 months, paralysis and/or dementia, unstable angina, history of myocardial infarction, congestive heart failure);
6. English-speaking and writing;
7. access and ability to use a computer for completion of online measures; and
8. possession of smartphone

Exclusion Criteria:

None

Ages: 19 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
change in OE importance, as measured by questionnaire | baseline 4- 8- and 12-weeks post intervention
change in OE accessibility, as measured by questionnaire | baseline 4- 8- and 12-weeks post intervention
change in OE certainty, as measured by questionnaire | baseline 4- 8- and 12-weeks post intervention

SECONDARY OUTCOMES:
change in intentions to exercise, as measured by questionnaire | baseline 4- 8- and 12-weeks post intervention
change in total weekly minutes of exercise | baseline 4- 8- and 12-weeks post intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University School of Nursing, Durham, North Carolina, United States